CLINICAL TRIAL: NCT02223715
Title: A Prospective Study to Characterize the Management and Outcome of Clostridium Difficile Infection （CDI) in Asian Pacific Countries
Brief Title: Prospective Observational Study of Clostridium Difficile Infection in Asian Pacific Countries
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 341-12-003
Record Dates: First submitted 2014-04-22; First posted 2014-08-22 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CDI
  Interventions: Other: CDI Pts

INTERVENTIONS:
Other: CDI Pts

SUMMARY:
The aim of this study is to conduct an Asia-Pacific, multi-center, prospective observational study to characterize patients with CDI as well as to understand treatment and management of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of CDI, as documented by diarrheal symptoms and positive stool test result for CDT or toxigenic C. difficile, or colonoscopic findings of PMC
* Patients and/or legal guardian willing to provide informed consent and/or informed assent or data release, according to local regulations

Exclusion Criteria:

* Patients with diarrheal symptoms caused by bacteria other than C. difficile, such as Salmonella, Campylobacter, Vibrio, Shigella, and Escherichia coli.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of CDI(C. difficile infection) who willing to provide informed consent and/or informed assent or data release, according to local regulation.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kanto Region, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Clostridium Difficile Infection: To characterize the ｍanagement and outcome of Clostridium Difficile Infection in asian pacific countries
Period: Overall Study
Arm/Group | Clostridium Difficile Infection
Started | 600
Completed | 496
Not Completed | 104
Not completed — Death | 31
Not completed — Lost to Follow-up | 73

BASELINE CHARACTERISTICS:
Groups:
- Clostridium Difficile Infection: Patient with Clostridium Difficile Infection
Arm/Group | Clostridium Difficile Infection
Number analyzed (Participants) | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 79
  Between 18 and 65 years | 241
  >=65 years | 280
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.0 [45.0 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272
  Male | 328
Region of Enrollment [Number; unit: participants]
  Japan | 48
  Australia | 60
  China | 64
  Hong Kong | 36
  India | 2
  Indonesia | 7
  Philippines | 9
  Singapore | 66
  Thailand | 44
  Vietnam | 64
  Malaysia | 2
  Korea, Republic of | 99
  Taiwan | 99

OUTCOME MEASURES:

1. Primary Outcome: Patient Demographics
Description: Medical history is information which was collected at the CDI diagnosis in this study. The items of the Medical history are indicated below. Concomitant diseases at the CDI diagnosis were included in the Medical history.
Time Frame: At the study at the time of CDI diagnosis enrollment
Population: Medical history is information which was collected at the CDI diagnosis in this study. The items of the Medical history are indicated below. Concomitant diseases at the CDI diagnosis were included in the Medical history.
Measure: Number; unit: participants
Groups:
- Medical History: To characterize the management and outcome of Clostridium Difficile Infection
Arm/Group | Medical History
Number analyzed (Participants) | 600
participants
  Myocardial infarction | 54
  Congestive heart failure | 46
  Cerebrovascular disease | 63
  Peripheral vascular disease | 29
  Chronic pulmonary disease | 57
  Connective tissue disease | 72
  Peptic ulcer disease | 69
  Liver disease | 76
  Diabetes mellitus | 154
  Renal disease | 143
  Solid tumor | 145
  Leukaemia | 44
  Lymphoma | 39
  AIDS | 3
  IBD | 68
  Nasogastric tube in past 30 days | 107
  Abdominal surgery in past 30 days | 36

2. Primary Outcome: Status at the End of CDI Episode
Description: The patients were observed from the diagnosis to the end of the treatment and got a telephone follow up call after two month from the end of treatment. The categories of the status indicating below are at the end of the treatment, not at the follow up call. Lost to follow-up means the patient number who were lost during the treatment course.
Time Frame: From the time of CDI diagnosis to the end of the treatment
Measure: Number; unit: participants
Groups:
- Status at the End of CDI Episode: To characterize the management and outcome of Clostridium Difficile Infection
Arm/Group | Status at the End of CDI Episode
Number analyzed (Participants) | 600
participants
  Lost to follow-up | 7
  Resolved | 562
  Death | 31

3. Secondary Outcome: Clinical Complication
Description: This study was non-interventional observational study. There were no restriction on the CDI treatment and we did not define to collect AE data. We just defined to collect the data for complications with CDI treatments indicating below. The complications to be checked were defined in the protocol. The information of other complications and AEs were not collected.
Time Frame: From the time of CDI diagnosis to recovery or recurrence
Measure: Number; unit: participants
Arm/Group | Clinical Complication
Number analyzed (Participants) | 600
participants
  Emergency colectomy performed | 2
  Colonoscopy/sigmoidoscopy performed | 2
  Colitis or PMC | 83
  Toxic megacolon | 1
  Hypokalaemia | 23
  Hypotension | 1
  Dehydration | 17
  Septic shock | 9
  Peritonitis | 4

4. Secondary Outcome: Recurrence or Not After 2 Months Follow-up
Description: The patients were observed from the diagnosis to the end of the treatment and got a telephone follow up call after two month from the end of treatment.
  Unknown includes patient lost, data missing
Time Frame: From the time of CDI diagnosis to 2 months follow-up
Measure: Number; unit: participants
Arm/Group | Recurrence or Not After 2 Months Follow-up
Number analyzed (Participants) | 600
participants
  Recurrence | 48
  No recurrence | 332
  Unknown | 220

ADVERSE EVENTS:
Description: Adverse Events were not pre-specified to be collected for this observational study. However, complications associated with CDI treatment were collected and are reported as an Outcome Measure.
Arm/Group | Clostridium Difficile Infection
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No